CLINICAL TRIAL: NCT00909493
Title: Nova Scotia Chronic Pain Collaborative Care Network: A Pilot Study
Brief Title: Chronic Pain Care Network
Acronym: NSCPCCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Anesthesiologists' Society (Other)
Responsible Party: Principal Investigator, Peter MacDougall, MD FRCPC, Nova Scotia Health Authority
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDHA-RS/2008-006
Record Dates: First submitted 2009-04-16; First posted 2009-05-28 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Pain
Keywords: Improvement of patient care as measured by self-rated health and improve physician satisfaction with chronic pain management
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Access to Pain Specialist (Experimental): Network
  Interventions: Other: Network Access

INTERVENTIONS:
Other: Network Access — Primary Care Physicians in this treatment group will have access to a pain specialist at the Pain Management Unit.

SUMMARY:
The proposed Nova Scotia Chronic Pain Collaborative Care Network (NSCPCCN) is a professional development partnership between family physicians and chronic pain and addiction specialists designed to build capacity in the health care system and provide improved pain management to patients. The NSCPCCN will provide community physicians with access to chronic pain and addiction specialists to assist in the management of patients with chronic pain. The current project is designed as a pilot project to determine the feasibility of a this program on a large scale. In order to determine the effect of implementation of a mentor- mentee network in the primary care setting, a pilot project will be undertaken. The study will assess the impact of the NSCPCCN on treatment of chronic pain and opiate management in two communities in Nova Scotia prior to a proposed province wide rollout of the program.

DETAILED DESCRIPTION:
Chronic pain is recognized as a world-wide problem. Gureje et al (1) demonstrated that 21% of patients presenting for primary care reported persistent pain and were four times more likely to have a depressive disorder than those without pain. One third of patients with persistent pain had a moderate to severe work role impairment (1). Canadian studies have demonstrated that up to 30% of the population suffers from chronic pain (2, 3). By extrapolation it may be expected that between 20-30% of persons living in Nova Scotia suffer from chronic pain.

Chronic pain is associated with significant morbidity and mortality. It is also associated with increased rates of depression, poorer self related health and increased risk of suicidality (2-4). Poor self-rated health has been demonstrated to be a predictor of increased morbidity and mortality (5-7). Tang and Crane (4) demonstrated that persons with chronic pain have a risk of death by suicide twice that of controls and that the lifetime prevalence of suicide attempts was 5-14%. Chronic pain impairs sleep (8) and may be related to abnormal immune function (9-11). As well, there is morbidity and mortality associated with medications used in the treatment of chronic pain. Although opiate medications form a significant part of the pain management armamentarium they are also associated with serious morbidity including sedation, respiratory depression, death and addiction. Death rates from these medications have risen dramatically (12) in recent years. Ives et al (13) report a 32% incidence of opiate misuse in an academic pain management unit. Cicero et al (14) reported that prescription opiate misuse is more common in rural, suburban and small urban areas, similar to the geographic background of Nova Scotia, and concluded that regionally specific risk minimization strategies should be developed.

The proposed Nova Scotia Chronic Pain Collaborative Care Network (NSCPCCN) is a professional development partnership between family physicians and chronic pain and addiction specialists designed to build capacity in the health care system and provide improved pain management to patients. The NSCPCCN will provide community physicians with access to chronic pain and addiction specialists to assist in the management of patients with chronic pain. The current project is designed as a pilot project to determine the feasibility of this program on a large scale. In order to determine the effect of implementation of a mentor- mentee network in the primary care setting, a pilot project will be undertaken to determine the feasibility and logistics of the NSCPCCN.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Physicians in Nova Scotia DHA 1

Exclusion Criteria:

* Primary Care Physicians outside of Nova Scotia DHA 1

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome for patients will be an improvement in self-rated health. | 9 months
The primary outcome for physicians will be an improvement in satisfaction in ability to manage chronic pain conditions. | 9 months